CLINICAL TRIAL: NCT04933149
Title: Ketamine Infusion for Treatment of Chronic Neuropathic Pain in Traumatic Brachial Plexus Injuries, a Prospective Randomized Control Study
Brief Title: Ketamine Infusion for Neuropathic Pain in Brachial Plexus Injuries
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Alexander Y. Shin, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-011213
Record Dates: First submitted 2021-06-15; First posted 2021-06-21 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Brachial Plexus Injury
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine Infusion Group (Experimental): Subjects will receive ketamine infusion during their planned surgery and postoperatively.
  Interventions: Drug: Ketamine Infustion
- Standard of Care Group (No Intervention): Subjects will receive general anesthesia as standard of care during their planned surgery

INTERVENTIONS:
Drug: Ketamine Infustion — Intravenous infusion at 0.5 mg/kg/hr from induction to emergence from anesthesia during the subject's brachial plexus reconstruction surgery. In addition, subjects will receive postoperative ketamine infusion of 0.1-0.3 mg/kg/hr for 24 hours titrated to side effects while patients are admitted to the hospital following surgery.
  Other Names: Ketamine
  Arms: Ketamine Infusion Group

SUMMARY:
The purpose of this study is to assess pre- and postoperative neuropathic pain in patients with traumatic brachial plexus injuries to determine if intraoperative ketamine infusion affect neuropathic pain associated with avulsion injuries of the brachial plexus.

DETAILED DESCRIPTION:
Neuropathic pain following traumatic brachial plexus injuries is a common and debilitating problem that has been reported in up to 64-75% of patients. Neuropathic pain is difficult to treat, particularly when secondary to avulsion injuries of the brachial plexus. Current treatment options include neuromodulating pharmacologic agents including gabapentin, pregabalin, tricyclic antidepressants, and duloxetine among others. Other analgesic modalities include TENS unit application, massage, acupuncture, and topical medications. Despite these treatment options, patients frequently continue to experience significant, debilitating neuropathic pain.

The use of ketamine has recently been studied in complex regional pain syndrome (CRPS), spinal cord injuries, and chronic neuropathic pain with encouraging results. Ketamine is thought to exert its analgesic properties via noncompetitive central nervous system N-methyl-D-aspartate (NMDA) antagonism among other primarily central mechanisms including sodium channel blockade, activation of D2 dopamine receptors and facilitation of γ-aminobutyric acid A (GABA-A) signaling. It is utilized clinically in acute and chronic pain management primarily in hospitalized settings to treat a variety of pain states as well as medically refractory depression and headache disorders. The dosing and administration of ketamine infusion varies widely across studies and includes oral ketamine, low dose infusions, and infusions producing an anesthetic effect. To our knowledge, ketamine's use in subanesthetic doses has not been adequately evaluated in patients with neuropathic pain following traumatic brachial plexus injuries. Our study aims to determine how intraoperative ketamine infusion alters neuropathic pain severity associated with brachial plexus avulsion injury in the post-operative period. In addition, we hypothesize that patients receiving intraoperative ketamine infusion will require less narcotic pain medication through the follow-up period of 6 months following surgery.

Patients who are undergoing planned surgery for brachial plexus reconstruction at Mayo Clinic will be enrolled into this study to be randomized into getting ketamine infusions or a placebo medication during surgery and in the 24 hour postoperative period after surgery. Pain will be measured before surgery and at various time points to up to 6 months after surgery through online pain measurement scores.

ELIGIBILITY:
Inclusion Criteria:

* Patients with neuropathic pain associated with avulsion injuries following traumatic brachial plexus injuries scheduled for brachial plexus exploration and reconstruction by three senior surgeons at Mayo Clinic (AYS, ATB, RJS):
* Neuropathic pain defined as pain directly related to injury to the somatosensory system, and score >4/10 on the Douleur Neuropathique en 4 Questions (DN4) neuropathic pain questionnaire. Symptoms of neuropathic pain include allodynia, hyperalgesia, burning, needle-like, throbbing, shooting, or electrical-type sensation.
* Nerve root avulsion on CT myelogram.
* Traumatic brachial plexus injuries defined as blunt or penetrating trauma resulting in injury and dysfunction along the course of the brachial plexus defined as nerve roots C5-T1, trunks, divisions, cords, and terminal branches.

Exclusion Criteria:

* Patients without pain following traumatic brachial plexus injuries.
* Patients with brachial plexus injuries due to non-traumatic causes such as tumors, infection, radiation, or inflammatory disorders such as Parsonage Turner Syndrome.
* Patients who do not require surgery for exploration/reconstruction at the brachial plexus.
* Patients under 18 years of age.
* Contraindication to ketamine use (severe hepatic dysfunction -cirrhosis, high-risk coronary artery disease, poorly controlled psychiatric condition- schizophrenia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in PROMIS Pain Quality - Neuropathic Pain (PQ-Neuro) score | Baseline, 1 week
  Measured by the PROMIS Pain Quality - Neuropathic Pain (PQ-Neuro) self-reported questionnaire asking about pain in the past 7 days using a scale of 1=not at all and 5=very much. Higher scores indicate a worse outcome.

SECONDARY OUTCOMES:
Opioid medication use | Baseline, 1 week postoperatively
  Change in opioid medication use measured by oral morphine equivalents (OMEs) at postoperative week 1 from baseline
Pain Score | 1 day postoperatively
  Measured using the Visual Analogue Scale for pain rated from 0-10, where 0 is no pain and 10 is the worst pain imaginable.
Adverse Events | 6 weeks
  Number of participants to experience sepsis, embolism, wound healing failure, hematomas, or nightmares/hallucinations following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Shin, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials